CLINICAL TRIAL: NCT01683526
Title: Safety and Efficacy of Endotracheal Intubation by Pulmonary Critical Care Physicians in Critically-Ill Patients Using Glidescope Video-Laryngoscope
Brief Title: Safety and Efficacy of Endotracheal Intubation Using Glidescope Video-Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 139-12
Record Dates: First submitted 2012-09-06; First posted 2012-09-12 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Respiratory Failure
Keywords: Urgent endotrachel intubation; Direct laryngoscopy; Video laryngoscopy; Glidescope; Critical Care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct laryngoscopy (Active Comparator): Intubation will be done using direct laryngoscopy
  Interventions: Procedure: Direct laryngoscopy
- Video laryngoscopy (Active Comparator): Intubation will be done using video laryngoscopy
  Interventions: Device: Video laryngoscopy (Glidescope)

INTERVENTIONS:
Procedure: Direct laryngoscopy
  Other Names: standard laryngoscope
  Arms: Direct laryngoscopy
Device: Video laryngoscopy (Glidescope)
  Other Names: Glidescope Video Laryngoscope
  Arms: Video laryngoscopy

SUMMARY:
The safety and efficacy of a video-laryngoscope as a primary intubation tool in urgent endotracheal intubation of critically-ill patients has not been well-described in the literature. This study will answer whether using a VL will impact on the efficacy and safety of intubation compared with a traditional direct laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing urgent endotracheal intubation by a pulmonary critical care medicine physician

Exclusion Criteria:

* Difficult airway
* Oxygen saturation < 92% despite adequate mask ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverberg, MD, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Isreal Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Direct Laryngoscopy: Intubation will be done using direct laryngoscopy
  Direct laryngoscopy
- Video Laryngoscopy: Intubation will be done using video laryngoscopy
  Video laryngoscopy (Glidescope)
Period: Overall Study
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Started | 60 | 57
Completed | 60 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (15.9) | 65.4 (14.0) | 67.4 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 56
  Male | 34 | 27 | 61

OUTCOME MEASURES:

1. Primary Outcome: First Pass Success Rate
Time Frame: From begining of intubation to verification. Less then 5 minutes approximatly
Measure: Number; unit: percentage of first pass success
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 60 | 57
percentage of first pass success | 24 | 42

2. Secondary Outcome: Severe Desaturation
Description: sat <80%
Time Frame: For 10 minutes post intubation
Measure: Number; unit: percentage of patients with desaturation
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 60 | 57
percentage of patients with desaturation | 5 | 2

3. Secondary Outcome: Hypotension
Description: SBP<70
Time Frame: For 10 minutes post intubation
Measure: Number; unit: percentage of hypotension
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 60 | 57
percentage of hypotension | 8 | 6

4. Secondary Outcome: Cardiac Arrest
Time Frame: For 1 hour post intubation
Measure: Number; unit: percentage of cardiac arrest
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 60 | 57
percentage of cardiac arrest | 0 | 1

5. Secondary Outcome: Complications of Intubation
Description: Complications of intubation including aspiration, vomiting, esophageal intubation,and dental injury.
Time Frame: For 10 minutes post intubation
Measure: Number; unit: percentage of other complications
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 60 | 57
percentage of other complications | 9 | 6

ADVERSE EVENTS:
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 0/60 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes